CLINICAL TRIAL: NCT00213291
Title: Extended Dosing of Darbepoetin Alfa (Aranesp) for the Management of Anemia in Children With Chronic Renal Failure
Brief Title: Darbepoetin Treatment of Anemia in Children With Chronic Renal Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Denis Geary, Nephrologist, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000004731
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Kidney Failure, Chronic
Keywords: chronic kidney failure; darbepoetin; pediatrics; anemia
MeSH Terms: conditions — Kidney Failure, Chronic; Anemia | interventions — Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: darbepoetin alfa

INTERVENTIONS:
Drug: darbepoetin alfa — Darbepoetin alfa will be administered by SC/IV injection every 14-28 days. Patients starting on the 14 day dose regimen will receive two times their baseline weekly dose; patients on the 28 day schedule will receive four times their average weekly dose. The exception to a Q14 or Q28 dosing schedule will be for patients requiring 10 mcg every 10 days. These patients will go to 20 mcg Q21 days before extending to the Q28 day schedule. Naive patients will start on a dose of 0.9 mcg/kg every 14 days. Study subjects who are successfully treated for 12 weeks on the 14 day schedule may be enrolled in the 28 day schedule study.

SUMMARY:
This is a study to determine the safety and effectiveness of Darbepoetin (Aranesp) given every 14 to 28 days to treat low red blood cells in children with chronic kidney failure.

DETAILED DESCRIPTION:
Erythropoietin (EPO) is a glycoprotein synthesized in the kidneys which regulates the rate of proliferation and differentiation of red blood cell precursors. The main cause of anemia in children with chronic renal failure is deficiency of EPO production as a result of declining renal function. Recombinant human EPO (rHuEPO) is a synthetic erythropoietin that is structurally and functionally similar to naturally occuring EPO. Treatment of anemia using rHuEPO has been associated with an improvement in the quality of life for patients, likely attributable to an increased production in hemoglobin and a reduction of dilatation of the heart. Recently, an analogue of EPO with two extra oligosaccharide chins, darbepoetin alfa, has been described as having a more prolonged effect requiring less frequent dosing.

There are currently no data available on the efficacy of darbepoetin alfa administered every 14-28 days for children. The most common dosing schedules in the clinical trial at HSC are every 7, 10, and 14 days. Due to reports of increased pain associated with the SC injection, and confusion of caregivers when the 10 day dosing schedule is necessary, the goals of the current proposal are to: 1) Decrease the frequency of SC injections and 2)Eliminate the 10 day dosing schedule for the administration of Darbepoetin.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic renal insufficiency or end stage renal disease (ESRD) requiring dialysis
* clinically stable
* hemoglobin of 110-125 g/L in screening period; for naive subjects, hemoglobin < 110 g/L
* not iron deficient (TSAT > 19.5%) within 4 weeks of study entry
* stable darbepoetin alpha therapy administered IV or SC q7 to q21 days OR darbepoetin alpha naive
* written informed consent from parent/legal guardian
* less than 18 years old
* weight at least 10 kg
* females of childbearing potential must practice adequate contraception
* availability for follow-up assessments

Exclusion Criteria:

* scheduled for a living donor kidney transplant within 12 weeks of signing consent
* uncontrolled blood pressure as judged by principal investigator
* change in seizure pattern in past 30 days; grand-mal seizure 12 weeks before enrollment
* current clinical evidence of severe hyperparathyroidism
* major surgery 2 weeks before signing consent
* active inflammatory disease or condition requiring immunosuppressive therapy
* currently receiving antibiotics for active systemic infection
* peritoneal dialysis patient with an episode of peritonitis within the past 30 days
* known HIV antibody positivity
* known antibodies to rHuEPO
* known aluminum toxicity
* known red cell aplasia
* known malignancy

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2005-04; Primary Completion 2005-09 (Actual); Study Completion 2005-10

PRIMARY OUTCOMES:
The safety of darbepoetin when administered at an increased dosing interval | 40 weeks

SECONDARY OUTCOMES:
Safety and tolerability of darbepoetin | 40 weeks
Proportion of subjects who receive red blood cell transfusions | 40 weeks
Percentage of Hb data points that exceed upper target of 125 g/L | 16-36 weeks
Incidence of anti-erythropoietin antibody formation | 40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Denis F Geary, MD, Principal Investigator — The Hospital For Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada